CLINICAL TRIAL: NCT06716905
Title: A Single-Center, Randomized, Double-Blind, Placebo-Controlled, Phase I Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Dose Escalations of ACT500 (Formerly Known as NM6606) in Chinese Healthy Adult Participants
Brief Title: Safety, Tolerability, and Pharmacokinetics of ACT500 in Healthy Adult Participants
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xiamen Amoytop Biotech Co., Ltd. (Industry)
Collaborators: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ACT500-4/01
Record Dates: First submitted 2024-11-13; First posted 2024-12-04 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Non-alcoholic Steatohepatitis
Keywords: Non-alcoholic Steatohepatitis; ACT500; NM6606; pharmacokinetic
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1:ACT500 Tablets (Experimental)
  Interventions: Drug: ACT500 tablets
- Part 1: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Part 2:ACT500 Tablets (Experimental)
  Interventions: Drug: ACT500 tablets
- Part 2: Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ACT500 tablets — Participants will receive a single ascending oral dose of ACT500 Tablets under fasting state on the first day in Part 1
  Arms: Part 1:ACT500 Tablets
Drug: Placebo — Participants will receive placebo matched to ACT500 Tablets.
  Arms: Part 1: Placebo
Drug: ACT500 tablets — Participants will receive multiple ascending oral dose of ACT500 Tablets under fasting state once daily for 7 days in Part 2.
  Arms: Part 2:ACT500 Tablets
Drug: Placebo — Participants will receive placebo matched to ACT500 Tablets.
  Arms: Part 2: Placebo

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled Phase I clinical study, divided into two parts. The first part is a single-dose escalation study (Part1,SAD study phase), and the second part is a multiple-dose escalation study (Part2,MAD study phase). It's aimed to evaluate the safety, tolerability, and pharmacokinetics (PK) of ACT500 in healthy adult participants, and to explore possible metabolites and biomarkers of ACT500.

ELIGIBILITY:
Inclusion Criteria:

* Participants are willing and able to sign a written informed consent form voluntarily before starting any study-related procedures and are willing to comply with all required study procedures;
* Males or females between 18 and 55 years of age (inclusive) at the time of screening;
* Body Mass Index (BMI) between 19-26 kg/m^2 (inclusive) at the time of screening, with a weight of at least 50 kg;
* Blood pressure within the normal range at the time of screening: systolic pressure: 90-139 mmHg, diastolic pressure: 60-89 mmHg (inclusive of the critical values);
* Participants of men and women of childbearing potential willing to use highly effective contraceptive measures (condoms, contraceptive sponges, contraceptive gels, contraceptive films, intrauterine devices, oral or injectable contraceptives, subdermal implants, etc.) from the time of signatures of the informed consent form until 90 days after the last administration of the study medication; and women of childbearing potential must have a negative serum pregnancy tests at the time of screening and at the time of the D-1 examination;

Exclusion Criteria:

* Allergic to the study drug or any of its components;
* Have previously used the study drug;
* Have clinically significant diseases, including but not limited to abnormality in liver or kidney, blood, digestive (including bleeding, infection, obstruction, or diarrhea greater than grade 1), respiratory, cardiovascular and cerebrovascular, endocrine, metabolic disorders, nervous system diseases, etc., which assessed by the investigator unsuitable for inclusion;
* Clinical significant abnormality in vital signs, physical examination, laboratory tests, or ECG at screening, as assessed by the investigator unsuitable for inclusion;
* QTcF > 450ms (males), QTcF > 480ms (females) at screening [Fridericia's formula: QTcF = QT/(RR)^1/3];
* Estimated glomerular filtration rate (eGFR) < 90 mL/min/1.73m^2 at screening;
* A history of unstable cardiovascular and cerebrovascular diseases within 6 months prior to screening, including acute myocardial infarction, stroke, arrhythmia, etc.;
* Existing liver disease or unexplained elevation of liver function tests (alanine aminotransferase (ALT), aspartate aminotransferase (AST), gamma-glutamyl transferase (GGT), alkaline phosphatase (ALP), total bilirubin or direct bilirubin > 1.5×ULN at screening or D-1, or D-1 test value is more than 50% higher than the screening test value);
* Respiratory infections (upper and/or lower respiratory tract) treated with antibiotics within 12 weeks before screening;
* Infectious diseases within the screening period (within 28 days before the first dose) that, in the investigator's judgment, would affect the participant's ability to participate in the trial;
* History of tuberculosis;
* History of malignant tumors (except for basal cell carcinoma or squamous cell carcinoma of the skin);
* Serious trauma or surgery within 28 days before the first dose, or planning major surgery during the study period;
* Blood donation or significant blood loss (≥400mL) within 56 days before the first dose, or having received a blood transfusion;
* Use of any medication (including prescription drugs, over-the-counter drugs, traditional Chinese medicine, etc.) or health products within 14 days before the first dose (or 5 half-lives, whichever is longer);
* Use of strong inhibitors or inducers of CYP450 enzymes and/or P-gp within 28 days before the first dose, or needing to continue using the above drugs during the study period;
* Received live or attenuated vaccines within 30 days before the first dose, or planning to receive them during the study period;
* Participated in or currently participating in other new drug or medical device clinical trials within 30 days before the first dose (or 5 half-lives, whichever is longer), or currently undergoing follow-up of another clinical study;
* Unable to swallow oral medication, having clinically significant gastrointestinal abnormalities (such as post-gastrointestinal resection, post-gastrointestinal anastomosis, chronic diarrhea, and intestinal obstruction, etc.) or existing conditions that, in the investigator's judgment, significantly affect gastrointestinal absorption;
* Poor venous access, unable to tolerate venipuncture, or having a history of clinically significant syncope or needle phobia as judged by the investigator;
* History of drug or substance abuse;
* Positive results for any of the following tests during the screening period: human immunodeficiency virus antibody (HIV-Ab), syphilis antibody, hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV-Ab);
* Heavy smoking (defined as more than 5 cigarettes per day) or use of nicotine-containing products (such as snuff, nicotine patches, nicotine gum, e-cigarettes, simulated cigarettes, or inhalers) within 6 months before screening; or unable to quit smoking (stop nicotine intake) during the trial period;
* A history of alcohol abuse within 90 days before screening, or positive alcohol test results at D-1; or unable to abstain from alcohol intake during the trial period; alcohol abuse is defined as an average weekly intake of more than 14 standard drinks (1 standard drink contains 14g of alcohol, such as 45ml of spirits with an alcohol concentration of 40% or 180ml of wine with an alcohol concentration of 10%);
* Pregnant or breastfeeding women;
* The investigator believes that the participant has other conditions that may affect compliance or are unsuitable for participation in this trial.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-03-06 (Actual); Primary Completion 2025-09-22 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Event（AE） | SAD:Day1-8; MAD:Day1-22.
Serious Adverse Event | SAD:Day1-8; MAD:Day1-22.
body temperature | SAD:Day1-5; MAD:Day1,Day7-22.
respiration | SAD:Day1-5; MAD:Day1,Day7-22.
pulse | SAD:Day1-5; MAD:Day1,Day7-22.
heart rate | SAD:Day1-5; MAD:Day1,Day7-22.
blood pressure | SAD:Day1-5; MAD:Day1,Day7-22.
Physical Examination | SAD:Day1,Day3-8; MAD:Day1,Day3-22.
  Physical examination includes general condition, head and neck, lymph nodes, skin, chest, abdomen, and musculoskeletal system (including limbs and spine).
Number of Participants with 12-Lead Electrocardiogram Findings | SAD:Day-1,Day5 ; MAD:Day-1,Day3,Day8and D14.
Number of Participants with Dynamic electrocardiogram（ECG）Findings | SAD:Day1; MAD:Day1,Day7.
Number of Participants with Abnormal Laboratory Parameters Findings | SAD:Day1-8; MAD:Day1-22.

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | SAD:Day1-5;
Time to maximum concentration(Tmax) | SAD:Day1-5;MAD:Day1-8
The area under the plasma concentration-time curve from the time of initial dosing to the time of the last measurable concentration point (AUC0-t) | SAD:Day1-5;
The area under the plasma concentration-time curve from the time of initial dosing to infinity (AUC0-∞) | SAD:Day1-5;
Apparent terminal elimination half-life (t1/2). | SAD:Day1-5;
Clearance (CL/F) | SAD:Day1-5;
Apparent Volume of Distribution (Vd/F) | SAD:Day1-5;
Elimination Rate Constant（Kel） | SAD:Day1-5;
Mean Residence Time（MRT） | SAD:Day1-5;
Steady-state trough concentration(Cmin,ss) | MAD:Day1-8;
Steady-state peak concentration(Cmax,ss) | MAD:Day1-8;
Average steady-state plasma concentration(Cav,ss) | MAD:Day1-8;
Elimination half-life(t1/2,ss) | MAD:Day1-8;
Clearance (CLss/F) | MAD:Day1-8;
Apparent Volume of Distribution (Vd/Fss) | MAD:Day1-8;
Accumulation Index (RAC) | MAD:Day1-8;
The area under the plasma concentration-time curve from the time of the last dose to the time of the last measurable concentration point (AUC0-t,ss) | MAD:Day1-8;
The area under the plasma concentration-time curve within one dosing interval after the last dose (AUC0-τ) | MAD:Day1-8;
The area under the plasma concentration-time curve extrapolated from the last dose to infinity (AUC0-∞,ss) | MAD:Day1-8;
Coefficient of Fluctuation (DF) | MAD:Day1-8;
Pharmacokinetic (PK):Plasma Concentrations of ACT500 | SAD:Day1-4;MAD:Day1-8;
Changes of biomarkers after single and multiple oral dosing compared to baseline | SAD:Day1-5;MAD:Day1-8.

CONTACTS AND LOCATIONS:
Overall Officials: JianYing Huang, Principal Investigator — Zhongnan Hospital
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No